CLINICAL TRIAL: NCT03864731
Title: Audiological Benefit and Improved Quality of Life in Patients With a Bone Conduction Device - a Randomized Controlled Trial
Brief Title: Quality of Life With Bone Conduction Hearing Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Valerie Dahm, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2087/2018
Record Dates: First submitted 2019-02-24; First posted 2019-03-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Conductive Hearing Loss
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone conduction device - ADHEAR (Other): Patients will receive a hearing aid (ADHEAR). Hearing assessment will be carried out. Quality of life measurement will be carried out.
  Interventions: Device: Bone conduction device (ADHEAR)

INTERVENTIONS:
Device: Bone conduction device (ADHEAR) — adhesive bone conduction device

SUMMARY:
The aim of this study is to compare the audiological and quality of life performance patients have with an ADHEAR (adhesive bone conduction device) compared to no hearing device.

DETAILED DESCRIPTION:
Patients will be recruited at the outpatient's department of the Medical University of Vienna - Otorhinolaryngology department. Patient will be asked to participate in the study when inclusion and exclusion criteria are met. Mostly patients scheduled for a surgery improving conductive hearing loss or scheduled for implantation of an implantable bone conduction hearing aid will be included in the study.

Patients who do not use a hearing aid and who are not planning on using a hearing aid meeting the inclusion and exclusion criteria will also be asked to participate in the study. After inclusion in the study patients will be asked to fill out two questionnaires (quality of life and hearing specific questionnaire). They will then be fitted with an ADHEAR device and undergo unaided and aided soundfield audiometry. Randomization will be carried out (Randomization ratio 1.4:1) and patients in the intervention group will keep the device for the following 4 months with one visit after the first probation time of one month. At the one month mark patients in the control group will be asked to fill out the two questionnaires. Patients in the control group will be asked to return to the department and fill out the three questionnaires (SSQ-12 (Speech Spatial and Hearing Questionnaire), AQoL(Assessment of Quality of Life) and In-house questionnaire). Further audiologic assessment will be carried out. At this appointment patients will be able to talk about their experiences in the probation period und easily terminate the study in case of insufficient improvement, pain, skin irritations or other issues. At the four month mark patients in both groups will be asked to return for audiologic assessment and for filling out the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral and/or bilateral conductive hearing loss (CHL)
* Conductive hearing loss >10 decibel on average
* Subjective benefit from the device
* Subjects aged 13 years or older
* Capable of the German language
* Willingness and ability to perform all tests required for the study
* Signed, and dated informed consent before the start of any study specific procedure

Exclusion Criteria:

* Pregnancy or breastfeeding
* Patient uses a hearing aid or plans to acquire a hearing aid
* Patient is intolerant of the materials as described by Manufacturer
* Patient presents with a skin or scalp condition that may preclude the attachment of the adhesive adapter.
* Patient cannot perform the audiological tests or is unable to fill out the questionnaires.
* Patient presents with retrocochlear, or central auditory disorder.
* any physical, psychological, or emotional disorder that would interfere with the ability to perform on test and rehabilitation procedures

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
AQoL (Assessment of Quality of Life) Results | 4 months
  The primary objective of this study is to evaluate, whether patients using ADHEAR have a significantly improved quality of life compared to patients not fitted with a device with the AQoL (Assessment of Quality of Life) questionnaire. It comprises 35 questions covering a multitude of quality of life aspects. Weighted utilities are generated using the algorithms provided on the AQoL website. Weighted utilities give a number between 0 and 1 as answer for every question. These sub scores are then presented.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Dahm, MD, Principal Investigator — MUW
Locations (1):
- MUW AKH, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No